CLINICAL TRIAL: NCT05956171
Title: The Effects of Two Different Treatment Protocols on Shoulder Function, Quality of Life, and Ultrasound Parameters in Patients With Frozen Shoulder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Fatmanur Yegin, Research Assistant Doctor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/890
Record Dates: First submitted 2023-07-14; First posted 2023-07-21 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Frozen Shoulder; Shoulder Capsulitis; Shoulder Pain
Keywords: hydrodilatation; hydrodistension; ultrasound
MeSH Terms: conditions — Bursitis; Shoulder Pain | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: Two-arm study with one hydrodilatation group compared with the standart treatment group(cortisteroid injection)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound Guided Hydrodilatation with corticosteroid injection (Experimental): 15 ml intra-articular injection to shoulder via anterior approach under ultrasound guidance
  Drugs:
  * betamethasone dipropionate/ betamethasone sodium phosphate(diprospan) (5 mg+2mg/ml) (1 ml)
  * prilocaine hydrochloride %2 (4 ml)
  * Sodium chloride %0,9 (10 ml)
  Interventions: Other: Ultrasound Guided Hydrodilatation with corticosteroid injection
- Blind intra-articular corticosteroid injection (Active Comparator): 5 ml intra-articular blind injection to shoulder via posterior approach
  Drugs:
  * betamethasone dipropionate/ betamethasone sodium phosphate(diprospan) (5 mg+2mg/ml) (1 ml)
  * prilocaine hydrochloride %2 (4 ml)
  Interventions: Other: Intra-articular corticosteroid injection

INTERVENTIONS:
Other: Intra-articular corticosteroid injection — 5 ml blind intra-articular corticosteroid injection
  Arms: Blind intra-articular corticosteroid injection
Other: Ultrasound Guided Hydrodilatation with corticosteroid injection — 15 ml intra-articular injection to shoulder via anterior approach under ultrasound guidance
  Arms: Ultrasound Guided Hydrodilatation with corticosteroid injection

SUMMARY:
The goal of this interventional study is to compare the outcomes of two different injection aprroaches in patients with frozen shoulder. The main questions it aims to answer are:

* Is hydrodilatation better than intraarticular corticosteroid injection?
* Is there any prognostic factors that will help clinicians guide their decision making when choosing between these two treatments?

Participans will receive an injection(cortcosteroid and local anesthetics alone or with hydrodilatation-corticosteroid and local anesthetics plus sterile saline solution) and then they will follow a rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Patients who fulfill the diagnostic criteria for frozen shoulder
* Agree to participate in the study
* Having the opportunity to follow up for at least 3 months

Exclusion Criteria:

* Refusing to participate in the study
* History of shoulder injection in the last 3 months
* Having diabetes mellitus
* Presence of comorbidities that contraindicate injection therapy, such as bleeding diathesis
* Known history of allergy or anaphylaxis to drugs used in treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline pain score on Visual Analog Scale(VAS) | Baseline, 1 week, 1 month, 3 months
  Pain scored according to VAS; between 0(no pain) to 10(worst pain)
Change in Shoulder Pain and Disability Index(SPADI) scores | Baseline, 1 month, 3 months
  Scored between 0-10 ; 0 means no pain and disability and 10 means the worst pain and disability

SECONDARY OUTCOMES:
Change in Range of Movement(ROM) | Baseline, 1 week, 1 month, 3 months
  Range of shoulder movements assessed with digital inclinometer in sittting and lying positions
Ultrasound Parameters | Baseline, 1 month, 3 months
  Coracohumeral ligament(CHL) thickness, axillary pouch(AP) thickness, elastography of deltoid muscle(anterior, middle, and posterior)
Proprioception(Active position sense- joint position error) | Baseline, 3 months
  Shoulder joint is positioned in 30 degree flexion and 15 degree internal and external rotation in lying position, patient is asked to position their joints and errors in degrees noted
Shoulder Strength | Baseline, 3 months
  Measured with cybex isokinetic dinamometer, shoulder flexion/extension and shoulder internal/external rotation
Changes in Depression Score | Baseline, 1 months, 3 months
  measured by Beck's Depression Inventory(between 0 to 40), 0 means no depression and 40 means severe depression
Changes in Life Quality Score | Baseline, 1 month, 3 months
  Items from the SF-36 (Short Form 36) survey, between 0(worst) to 100(best)
Treatment Satisfaction | 3 months
  Global Improvement and Satisfaction Score, between 1 to 5, 1 very dissatisfied, and 5 very satisfied

IPD SHARING:
Plan to Share IPD: No